CLINICAL TRIAL: NCT00831870
Title: PRessure and Imaging-Using the CardioMEMS EndoSure Sensor for Long-term Follow-up After EVAR With Standard Surveillance (Prospective Registry)
Brief Title: EndoSure Sensor for Long-term Follow-up After Endovascular AAA Repair
Acronym: PRICELESS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: CardioMEMS (Industry)
Responsible Party: Sponsor
Other Study IDs: CM-06-02b
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: EndoSure Sensor; s2 Sensor; abdominal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect and compare EndoSure and EndoSure s2 Wireless AAA Pressure Sensor measurements with measurements from CT scan imaging, ultrasound, and other tests used to measure your AAA sac size and endoleaks following AAA repair, and during follow-up visits with your physician. An antenna is held over the patient's abdomen to measure pressure inside the aneurysm sac. The reading does not cause any discomfort, and dye or radiation is not needed to take the pressure measurement. To qualify, the patient must have a previously implanted EndoSure Sensor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from subject or legal guardian
* Males or females, at least 18 years of age
* Subjects who are post-EndoSure Wireless AAA Pressure Sensor implantation, with pressure measurements at implant.
* Subjects willing to comply with the site-specific follow-up requirements of the investigator.

Exclusion Criteria:

* Subjects whose clinical condition, in the Investigator's opinion, would not allow them to complete participation in the registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female subjects, at least 18 years of age, who are post-EndoSure AAA Pressure Sensor implantation at time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2008-10; Study Completion 2012-10 (Estimated)